CLINICAL TRIAL: NCT03202758
Title: Phase Ib/II Trial Evaluating the Safety, Tolerability and Immunological Activity of Durvalumab (MEDI4736) (Anti-PD-L1) Plus Tremelimumab (Anti-CTLA-4) Combined With FOLFOX in Patients With Metastatic Colorectal Cancer
Brief Title: Evaluation of the Safety and the Tolerability of Durvalumab Plus Tremelimumab Combined With FOLFOX in mCRC
Acronym: MEDITREME
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDI-TREME-COLON
Record Dates: First submitted 2017-06-07; First posted 2017-06-29 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Durvalumab; Tremelimumab; FOLFOX; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — durvalumab; tremelimumab; Folfox protocol

STUDY DESIGN:
Intervention Model Description: Step 1: Phase Ib with the aim to confirmed the safety of the association of Durvalumab (q2w 750mg) + Tremelimumab (q4w 75mg) + FOLFOX
  Step 2: Phase II with the aim to assess efficacy of the association of Durvalumab (q2w 750mg) + Tremelimumab (q4w 75mg) + FOLFOX
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab + Tremelimumab + FOLFOX (Other): * Durvalumab for 12 months
  * Tremelimumab for up to 4 doses/cycles
  * FOLFOX
  Interventions: Drug: Durvalumab, Tremelimumab and ,FOLFOX

INTERVENTIONS:
Drug: Durvalumab, Tremelimumab and ,FOLFOX — Study will be performed in 2 step:
  STEP 1 (phase Ib) will assess the safety of the combination of Durvalumab 750mg q2w + tremelimumab 75mg q4w + FOLFOX during the 2 first cycles of treatment (1 month)
  STEP 2 (phase II) will assess the efficacy of the combination of Durvalumab 750mg q2w + tremelimumab 75mg q4w + FOLFOX

SUMMARY:
Colo-rectal cancer is still one of the leading causes of cancer death worldwide. In France, approximately 40 500 new cases are diagnosed each year. With more than 17 500 deaths in France in 2011, colo-rectal cancer is responsible for more than 12% of all cancer deaths, the overwhelming of deaths occurring in patients with metastatic disease.

Many studies highlight the fact that colo-rectal cancer has immunogenic properties and that host immune responses can influence survival. Recent data have provided a clearer understanding of the factors limiting the antitumor immune response in colo-rectal cancer. One of the most critical checkpoint pathways responsible for mediating tumor-induced immune suppression is the programmed death-1 (PD-1) and PD ligand 1 (PD-L1) pathway.

PD-1 is expressed on activated immune cells and can link to PD-L1 express on Antigen-Presenting-Cell. Usually, this pathway is involved in promoting T-cells tolerance and preventing tissue damage in settings of chronic inflammation. In pathological context, the PD-1/PD-L1 pathway contributes to immune suppression and evasion. Many human solid tumors including colo-rectal cancer express PD-L1, and this expression is associated with a worse prognosis. The interaction of PD-1 with the ligand PD-L1 inhibits T-cell proliferation, survival, and effectors functions; induces apoptosis of tumor-specific T cells; promotes the differentiation of CD4+ T cells into immunosuppressive regulatory T cells; and increases the resistance of tumor cells to cytotoxic T lymphocytes attack. Thus, the blockage of the PD-1/PD-L1 interactions represents a logical target for cancer immunotherapy and in particular colo rectal cancer immunotherapy strategy.

Preclinical studies have shown that PD-L1 blockade improves the immune response by restoring T-cell effectors functions. Recent work in two in vivo tumor models shows a strong interest in using an anti-PD-L1 in combination with standard treatment of colo-rectal cancer (FOLFOX). In these models, the survival of mice that are treated with the combination therapy reached 40% when no mice were alive with FOLFOX treatment alone. This result may be explained, in one hand by cytotoxicity of 5FU and in the other hand by the restoration of anti-tumor immune activity of anti-PD-L1. These results suggest that the combination of chemotherapy with immunotherapy would act synergistically in patients with colo-rectal cancer.

Research Hypothesis: Combination of chemotherapy (FOLFOX) with immunotherapy association (anti-PD-L1 + anti-CTLA-4) would act synergistically in patients with colo-rectal cancer.

DETAILED DESCRIPTION:
Phase Ib primary objective (STEP 1): To determine the safety of the combination of Durvalumab (Anti-PD-L1) + Tremelimumab (Anti-CTLA-4) + FOLFOX

Phase II primary objective (STEP 2): To determine the efficacy of the combination of Durvalumab (Anti-PD-L1) + Tremelimumab (Anti-CTLA-4) + FOLFOX in terms of progression free survival (PFS).

Phase II secondary Objective: To determine efficacy of the combination of Durvalumab (Anti-PD-L1) + Tremelimumab (Anti-CTLA-4) + FOLFOX in terms of response to treatment and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Male or female age more than 18 years
3. Performance status of 0 or 1 according to the ECOG and WHO
4. Histologically confirmed diagnoses of colorectal cancer with positive mutated KRas.
5. Patients with metastatic disease
6. First line therapy
7. Life expectancy of more than 12 weeks
8. Adequate normal organ and marrow function as defined below:

   * Haemoglobin > 9.0 g/dL
   * Absolute neutrophil count (ANC) > 1.5 x 109/L (>1500 per mm3)
   * Platelet count > 100 x 109/L (>100,000 per mm3)
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
   * Albumin > 30g/L
   * Creatinine < 1.5 X institutional upper limit of normal (ULN)
   * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
9. Tumour evaluation in the previous 4 weeks with presence of at least one measurable lesion according to RECIST 1.1 criteria
10. At least 4 weeks since the last chemotherapy, immunotherapy or other drug therapy and / or radiotherapy
11. Recovery to grade ≤ 1 from any AE derived from previous treatment according to the criteria of the NCI-CTCAE version 4.0
12. Biopsable disease (for ancillary studies) or willingness to provide consent for use of archieved tissue for research purposes
13. Female subjects must either be of non-reproductive potential or must have a negative serum pregnancy test upon study entry
14. Patients must be affiliated to a social security system
15. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site). Previous enrolment in the present study
2. Participation in another clinical study with an investigational product during the last 4 weeks
3. Any previous treatment with a PD-1 or PD-L1 /CTLA-4 inhibitor, including durvalumab or tremelimumab
4. History of another malignancy within the 5 previous years with low potential risk for recurrence other than :

   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ
5. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 28 days prior to the first dose of study drug (14 days prior to the first dose of study drug for subjects who have received prior TKIs (e.g., erlotinib, gefitinib and crizotinib) and within 6 weeks for nitrosourea or mitomycin C). (If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period may be required.)
6. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
7. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
8. Any history of hypersensitivity to durvalumab or tremelimumab, FOLFOX or their excipients
9. Any unresolved toxicity (CTCAE grade >1) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)
10. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
11. Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
12. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
13. History of primary immunodeficiency
14. History of organ transplant that requires use of immunosuppressive
15. History of allogeneic organ transplant
16. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection; Clinically significant cardiovascular disease including: myocardial infarction within 6 months,, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia; history of Mobitz II second degree or third degree heart block without a permanent pacemaker in place, hypotension; rest limb claudication or ischemia within 6 months; active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
17. Sever concurrent disease, or co-morbidity that in the judgment of the investigator, would make the patient inappropriate for enrolment
18. Ongoing treatment with CYP3A4 substrates or regularly taking of grapefruit juice
19. Known history of active tuberculosis
20. History of leptomeningeal carcinomatosis
21. Brain metastases or spinal cord compression
22. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
23. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
24. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
25. Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids
26. Subjects with uncontrolled seizures,
27. Subjects under guardianship, curatorship or judicial protection
28. Known allergy or hypersensitivity to IP or any excipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety of Durvalumab plus Tremelimumab in combination with FOLFOX chemotherapy | 1 month
  Criteria RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHRU Besançon, Besançon
  - Centre Georges François Leclerc, Dijon
  - CHU Nantes, Nantes
  - Hôpital Europeen Georges Pompidou, Paris
  - Hôpital Saint Antoine, Paris

REFERENCES:
- [Derived] Thibaudin M, Fumet JD, Chibaudel B, Bennouna J, Borg C, Martin-Babau J, Cohen R, Fonck M, Taieb J, Limagne E, Blanc J, Ballot E, Hampe L, Bon M, Daumoine S, Peroz M, Mananet H, Derangere V, Boidot R, Michaud HA, Laheurte C, Adotevi O, Bertaut A, Truntzer C, Ghiringhelli F. First-line durvalumab and tremelimumab with chemotherapy in RAS-mutated metastatic colorectal cancer: a phase 1b/2 trial. Nat Med. 2023 Aug;29(8):2087-2098. doi: 10.1038/s41591-023-02497-z. Epub 2023 Aug 10. PMID 37563240
- [Derived] Fumet JD, Isambert N, Hervieu A, Zanetta S, Guion JF, Hennequin A, Rederstorff E, Bertaut A, Ghiringhelli F. Phase Ib/II trial evaluating the safety, tolerability and immunological activity of durvalumab (MEDI4736) (anti-PD-L1) plus tremelimumab (anti-CTLA-4) combined with FOLFOX in patients with metastatic colorectal cancer. ESMO Open. 2018 Jun 19;3(4):e000375. doi: 10.1136/esmoopen-2018-000375. eCollection 2018. PMID 29942666